CLINICAL TRIAL: NCT00969670
Title: Correlation of Particulate Matter and Heme Oxygenase-1 Protein Activity in Asthmatic Children by Induced Sputum Analysis.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Elizabeth Fierman, PhD, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-09-LF-242-CTIL
Record Dates: First submitted 2009-08-29; First posted 2009-09-01 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Samples of indused sputum

SUMMARY:
Samples of sputum from asthmatic children, between 5-17 years, will be collected during two years of the study period to perform tests Particle Size Distribution (PSD) and Shape Analysis (SA) of the particulate matter in the sputum and a biochemical reaction to evaluate the activity of Heme Oxygenase-1 protein in sputum cell supernatants.

Each child will perform Pulmonary Function Testing (PFT) and Induced Sputum (IS) as a routine part of diagnosis of asthma.

Parents will be asked to complete a questionnaire including questions on their child's respiratory symptoms in the last 12 months as well as socioeconomic factors. Parents will be asked to give informed written consent for their child's participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* •All children, between 5-17 years, performing a routine diagnosis of asthma in Tel Aviv Sourasky Medical Center that there parents gave informed written consent for their child's participation in the study.

Exclusion Criteria:

* None.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children, between 5-17 years, performing a routine diagnosis of asthma in Tel Aviv Sourasky Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-10

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Laboratory of Tel Aviv Sourasky Medical Center, Tel Aviv, Israel